CLINICAL TRIAL: NCT03851107
Title: The Effectiveness of Participation-focused Interventions on Body Functions of Youth With Physical Disabilities: An Interrupted Time Series Design
Brief Title: The Effectiveness of Participation-focused Interventions on Body Functions of Youth With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Dana Anaby, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 151613
Record Dates: First submitted 2019-02-14; First posted 2019-02-22 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Cerebral Palsy; Spina Bifida; Muscular Dystrophies; Musculoskeletal Disorder
Keywords: participation; environmental barriers; youth; disabilities; body functions
MeSH Terms: conditions — Cerebral Palsy; Spinal Dysraphism; Muscular Dystrophies; Musculoskeletal Diseases | interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: An 18-week individual-based interrupted time series design with multiple baselines across 8 participants will be employed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based activity program (Experimental): Engagement in 6-week community-based activity program
  Interventions: Behavioral: Engagement in 6-week community-based activity program

INTERVENTIONS:
Behavioral: Engagement in 6-week community-based activity program — Participants engage in a 6-week community-based activity program of their choice. In order to engage in the selected activity, an Occupational Therapist (OT) will meet with each youth in their home. Using the PREP 5 steps (Make goals; Map out a plan; Make it happen; Measure the process and outcomes; Move forward) the youth will choose a community program. The OT will then search for the appropriate program, identify and remove potential environmental barriers for participation in that activity (e.g., accessibility, equipment) and educate program instructors regarding the youth's specific needs. This process, which includes up to 12 hours of working with the OT, will set the stage for enrolment of the youth in a community program for a period of 6 weeks - the actual intervention phase.
  Other Names: Pathways and Resources for Engagement and Participation

SUMMARY:
Youth with physical disabilities face greater restrictions to participation in community-based activities than their typically developing peers, which can lead to poor health outcomes. Emerging treatment approaches aimed at improving activity and participation have shifted from focusing only on impaired body functions towards the performance of functionally meaningful activities within the youth's natural environment. It is unclear, however, whether targeting intervention at the activity/participation level can, at the same time, result in improvement of personal functional skills (e.g., reaching) and body functions (e.g., range of motion) -components also important to address and maintain within the rehabilitation process. Together with key community-based stakeholders including youth/parents, clinicians, and policy-makers, the investigators plan, therefore, to examine whether engaging in a 6-week community based activity (e.g., joining a sledge hockey team, boccia) can lead to a significant improvement in three key body functions: motor, cognitive and affective functions. Eight participants with physical disabilities will take part in the study and engage in an activity program of their own choice. Changes in their body functions (e.g., movement-related functions, attention, behavior, mood) will be measured multiple times before, during and after the engagement in an individualized activity/program. Findings of this pilot study analyzed with input from key stakeholders can advance the investigators understanding about methods for testing complex and unique individual-based interventions. This can guide clinicians, families and policy-makers to select effective approaches that not only promote participation but can also facilitate additional (motor and mental) benefits from one single intervention. Such findings may also reduce the burdens on the healthcare system as well as on the youth and families.

DETAILED DESCRIPTION:
Youth with physical disabilities experience restrictions to participation in community-based activities, which can lead to poor health outcomes. Currently, activity-based treatment approaches that are client-centered and implemented in the youth's natural environment are considered recommended practice. It is unclear, however, whether targeting intervention at the activity and participation level (e.g. playing boccia) can result in improvement of body functions (e.g., joint mobility, balance) as well as in participation - two key outcomes of pediatric rehabilitation programs. Research suggests that the opportunity to practice therapist-prescribed exercise programs is positively associated with physical gains. However, the impact of participation in a chosen real-life activity that is meaningful to the youth on a range of body functions has not yet been established and effective methods for testing complex individual-based interventions and outcomes are lacking. With funding received from the Canadian Institutes of Health Research, the investigators have proven the effectiveness of the PREP intervention, i.e., Pathways and Resources for Engagement and Participation, in promoting youth participation in meaningful activities across two provinces. Using the PREP approach, the purpose of this pilot study is to 1) employ an interrupted time series (ITS) design in order to generate preliminary evidence on the effectiveness of participants engagement in a 6-week community-based activity program (e.g., team sledge hockey) on 3 body functions (i.e., motor, cognitive and affective) as well as on the performance of the selected activity. An 18-week interrupted time series design with multiple baselines across 8 participants with physical disabilities (e.g., cerebral palsy, spina bifida) will be employed. Each activity, individually selected by the participants, will be analyzed using the task analysis approach in order to identify the underlying body functions necessary for the chosen activity. These functions, i.e., motor (measured using the Spinal Alignment and Range of Motion Measure, the Functional Reach Test, the Trunk Impairment Scale and the Jamar dynamometer), cognitive and affective (using the Behavior Assessment System for Children), will then be measured multiple times throughout the entire study, resulting in overall 32 trajectories of change in body functions (8 participants X 3 body functions) and additional 8 trajectories representing change in activity performance (using the Canadian Occupational Performance Measure). Two experts will independently analyze each trajectory using visual inspection and an innovative analytical solution, i.e., a combination of segmented regression and mixed-effect modelling, will be performed to estimate the overall effectiveness of the intervention across participants. This interdisciplinary research team, including three researchers in the field of childhood disability (occupational therapy, physical therapy and pediatric medicine), has partnered with seven key stakeholders and will work collaboratively throughout the research process. This early study in the area will build knowledge about alternative clinical trials that can generate evidence applicable to practice. Findings can eventually inform decision-making by guiding clinicians, families and policy-makers in appraising the benefits of participation-based therapies on improving functional capacities and actual performance of meaningful life activities. Describing the multiple benefits potentially generated by one single intervention can facilitate the development of efficient youth-engaging therapies, and thereby contributing to the improvement of the provision of pediatric rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

* have a physical disability (e.g., cerebral palsy, spina bifida, musculoskeletal disorders, muscular dystrophy)
* restricted mobility, such as an inability to navigate all surfaces and stairs independently and safely without the use of aids, physical assistance or external support

Exclusion Criteria:

* Youth who are recovering within the first year following a severe brain injury or an orthopedic surgery will be excluded, as their functional capacities are less likely to be stable.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Anaby, PhD, Principal Investigator — McGill University
Locations (1):
- MAB-MACKAY Rehabilitation Center, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: To reach our sample size, we anticipated that there would be potential withdrawals. Hence, we approached 9 participants.
Groups:
- Community-based Activity Program: Engagement in 8-week community-based activity program
  Engagement in 8-week community-based activity program: Participants engage in a 8-week community-based activity program of their choice. In order to engage in the selected activity, an Occupational Therapist (OT) will meet with each youth in their home. Using the PREP 5 steps (Make goals; Map out a plan; Make it happen; Measure the process and outcomes; Move forward) the youth will choose a community program. The OT will then search for the appropriate program, identify and remove potential environmental barriers for participation in that activity (e.g., accessibility, equipment) and educate program instructors regarding the youth's specific needs. This process, which includes up to 12 hours of working with the OT, will set the stage for enrolment of the youth in a community program for a period of 8 weeks - the actual intervention phase.
Period: Overall Study
Arm/Group | Community-based Activity Program
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Community-based Activity Program: A 22-week individual-based interrupted time series design with multiple baselines was used (Clinical Trials identifier NCT03851107). The time-point in which the intervention, that is engagement in a chosen 8-week activity, was introduced varied. This resulted in different lengths of baselines, of 6 to 11 weeks, across participants.
Arm/Group | Community-based Activity Program
Number analyzed (Participants) | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 18 [17 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 7
Functional Issues [Mean (Full Range); unit: Number of checked items] — Functional issues are measured by a checklist that includes a list of 13 functional issues. The number of checked-off issues is counted and summed. The sum can range from 0 to 13. A higher number of functional issues indicate greater complexity of the youth's condition.
  Number of checked items | 3.7 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavioral Assessment System for Children
Description: The Behavioral Assessment System for Children, Third Edition is a valid and reliable 2-point and 4-point scale for evaluating 18 subscales of global mental and emotional functions. Subscales (e.g. anxiety, attention) include 7 to 13 items. T scores calculated using Pearson's Q-global testing system ranged from 0 to 120, with lower scores indicating higher cognitive and affective functions. Six subscales measuring attention problems, hyperactivity, anxiety, sense of inadequacy, self-esteem, somatization were measured. For each subscale, we plotted the repeated T scores and fitted it into a regression line to represent the average change across the 7 participants. We report the results of the two-level hierarchical models estimating the overall intervention effect size for each of the 6 cognitive and affective outcomes.
Time Frame: This outcome will be assessed repeatedly throughout the phases of the study of a period of 22 weeks: baseline (up to 11time-points; up to 11wks) intervention (8 time-points; 8wks) and follow-up (2-points, 4wks). A regression line fitted 22 observations.
Measure: Number (95% Confidence Interval); unit: fixed effects estimate
Groups:
- Change in Behavioural Assessment System for Children: Six subscales from the Behavioral Assessment System for Children (anxiety, attention problems, hyperactivity, self-esteem, somatization, sense of inadequacy) was measured repeatedly (weekly up to 22 weeks) throughout the phases of the study: baseline (up to 11time-points; up to 11 wks) intervention (8 time-points; 8 wks) and follow-up (2-points, 4 wks).
Arm/Group | Change in Behavioural Assessment System for Children
Number analyzed (Participants) | 7
fixed effects estimate
  Anxiety Subscale Baseline | 54.73 [41.91 to 67.55]
  Anxiety Subscale Change at Intervention | -3.35 [-7.82 to 1.11]
  Anxiety Subscale Intervention Trend | -0.05 [-0.40 to 0.30]
  Somatization Subscale Baseline | 64.38 [41.94 to 86.83]
  Somatization Subscale Change at Intervention | 0.69 [-2.68 to 4.07]
  Somatization Subscale Intervention trend | -0.01 [-0.30 to 0.28]
  Self-esteem Subscale Baseline | 62.89 [48.14 to 77.64]
  Self-esteem Subscale Change at intervention | -0.83 [-3.02 to 1.36]
  Self-esteem Subscale intervention trend | -0.03 [-0.27 to 0.21]
  Sense of inadequacy Subscale Baseline | 56.64 [47.18 to 66.11]
  Sense of inadequacy Subscale Change at intervention | -1.63 [-4.55 to 1.29]
  Sense of inadequacy Subscale Intervention trend | -0.11 [-0.50 to 0.28]
  Attention problems Subscale Baseline | 47.53 [40.27 to 54.80]
  Attention problems Subscale Change at intervention | -2.15 [-5.64 to 1.33]
  Attention problems Subscale Intervention trend | -0.30 [-0.59 to -0.01]
  Hyperactivity Subscale Baseline | 56.71 [51.77 to 61.64]
  Hyperactivity Subscale Change at intervention | -4.15 [-9.94 to 1.63]
  Hyperactivity Subscale Intervention trend | -0.49 [-0.95 to -0.02]

2. Primary Outcome: Change in Range of Motion Measure
Description: Measures motor body functions in terms of active/passive range of motion of lower and upper extremities. A score between 0 and 4 is calculated, with 4 being the most severe limitation in range of motion.
  The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.
Time Frame: This outcome will be assessed biweekly during the study (22 weeks): baseline (up to 6 time-points; up to 11wks) intervention (4 time-points; 8wks) and follow-up (1-point, 4wks). A regression line fitted all motor-related trajectories outcomes.
Measure: Count of Participants; unit: Participants
Groups:
- Change in Range of Motion Measure: Range of Motion was measured repeatedly (biweekly for up to 22 weeks) throughout the phases of the study: baseline (up to 6 time-points; up to 11 wks) intervention (4 time-points; 8 wks) and follow-up (1-point, 4 wks).
Arm/Group | Change in Range of Motion Measure
Number analyzed (Participants) | 7
Participants | NA — The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.

3. Primary Outcome: Change in Trunk Impairment Scale
Description: Assesses trunk control and includes 3 sub-scales; static sitting balance, dynamic sitting balance and coordination. It contains 17 items rated on a 2-, 3- or 4-point scale. Total score Measure motor body functions in terms of trunk control. Total score ranges from 0 (low performance) to 23 (high performance).
  The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Change in Trunk Impairment Scale: Trunk Impairment Scale was measured repeatedly (biweekly for up to 22 weeks) throughout the phases of the study: baseline (up to 6 time-points; up to 11 wks) intervention (4 time-points; 8 wks) and follow-up (1-point, 4 wks).
Arm/Group | Change in Trunk Impairment Scale
Number analyzed (Participants) | 7
Participants | NA — The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.

4. Primary Outcome: Change in Functional Reach Test
Description: Assesses motor body functions in terms of reaching. The maximum distance in inches the participant can reach forward while standing/sitting in a fixed position is measured: units: inches.
  The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Change in Functional Reach Test: Functional Reach Test was measured repeatedly (biweekly for up to 22 weeks) throughout the phases of the study: baseline (up to 6 time-points; up to 11 wks) intervention (4 time-points; 8 wks) and follow-up (1-point, 4 wks).
Arm/Group | Change in Functional Reach Test
Number analyzed (Participants) | 7
Participants | NA — The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.

5. Primary Outcome: Change in Jamar Dynamometer Strength Test
Description: Measures motor body functions in terns of maximal grip strength; units: pounds of force. Scores range from 0 to 200 pounds.
  The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Change in Jamar Dynamometer Strength Test: Jamar dynamometer strength test was measured repeatedly (biweekly for up to 22 weeks) throughout the phases of the study: baseline (up to 6 time-points; up to 11 wks) intervention (4 time-points; 8 wks) and follow-up (1-point, 4 wks).
Arm/Group | Change in Jamar Dynamometer Strength Test
Number analyzed (Participants) | 7
Participants | NA — The raw motor scores obtained from this assessment was not analyzed separately. Instead, we converted all the motor-related scores to standardized scores to create an index for motor measures. To describe the change observed more accurately we combined the trajectories of all motor scores into a regression line to represent the average change for all motor measures. The results of this analysis are presented in primary outcome 7.

6. Primary Outcome: Change in Canadian Occupational Performance Measure
Description: Canadian Occupational Performance Measure is a 10-point scale that measures activity performance. Score ranges from 1(unable to perform) to 10 (perform extremely well). A higher score represents higher perceived activity performance levels. A regression line was fitted to represent the average change for the 7 participants for performance (up to 22 observations).
Time Frame: This outcome will be assessed repeatedly throughout the phases of the study over a period of 18-weeks: baseline (8 time-points; 8 wks) intervention (6 time-points; 6 wks) and follow-up (2-points, 4 wks) resulting in a total of 16 data-points.
Measure: Number (95% Confidence Interval); unit: fixed effects estimate
Groups:
- Change in Canadian Occupational Performance Measure: Canadian Occupational Performance Measure was assessed repeatedly (weekly) throughout the phases of the study over a period of 18-weeks: baseline (11 time-points; 8 wks) intervention (8 time-points; 6 wks) and follow-up (2-points, 4 wks) resulting in a total of 22 data-points.
Arm/Group | Change in Canadian Occupational Performance Measure
Number analyzed (Participants) | 7
fixed effects estimate
  Canadian Occupational Performance Measure Baseline | 2.59 [1.83 to 3.36]
  Canadian Occupational Performance Measure Change at Intervention | 2.73 [0.81 to 4.65]
  Canadian Occupational Performance Measure Intervention trend | -0.49 [-0.95 to -0.02]

7. Primary Outcome: Change in Motor Outcomes
Description: Change in motor outcomes was determined by changes in scores (converted to standardized scores according to participant's baseline values) of range of motion (ROM), trunk impairment scale (TIS), functional reach test and Jamar dynamometer strength test (description of each outcome and its scores are presented in outcomes 2-5).
  We combined all motor-related trajectories outcomes into a regression line to represent the average change for all motor measures. A three-level hierarchical model was ﬁtted, with observations nested within outcomes nested within participants. The results of the combined trajectories are presented (rather than the raw motor scores) as they are more suited to describe the change observed.
Time Frame: This outcome will be assessed repeatedly throughout the phases of the study: baseline (up to 6 time-points; up to 11 wks) intervention (4 time-points; 8 wks) and follow-up (1-points, 4 wks; ).
Measure: Number (95% Confidence Interval); unit: fixed effects estimate
Groups:
- Change in Motor Outcomes: Changes in outcomes of range of motion (ROM), trunk impairment scale (TIS), functional reach test and Jamar dynamometer strength test were measured repeatedly (biweekly for up to 22 weeks) throughout the phases of the study: baseline (up to 6 time-points; up to 11 wks) intervention (4 time-points; 8 wks) and follow-up (1-point, 4 wks).
Arm/Group | Change in Motor Outcomes
Number analyzed (Participants) | 6
fixed effects estimate
  Combined intervention effect | 3.71 [-0.25 to 7.66]
  Change at intervention | 1.57 [-0.69 to 3.83]
  Intervention trend | 0.26 [0.03 to 0.49]

ADVERSE EVENTS:
Description: Given that this study is considered low-risk, all-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not assessed in a standardized manner and adverse events data were not collected.
Arm/Group | Community-based Activity Program
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03851107/Prot_SAP_000.pdf